CLINICAL TRIAL: NCT02970422
Title: COPD Patient Preferences, Activities, and Participation Survey
Brief Title: Chronic Obstructive Pulmonary Disease Patient Preferences Survey
Status: Completed | Type: Observational
Sponsor: McGill University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Dennis Jensen, Ph.D., Assistant Professor, McGill University
Other Study IDs: 15-203-MUHC
Record Dates: First submitted 2016-04-26; First posted 2016-11-22 (Estimated); Results first posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Survey; Priorities; Activities; Participation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Quartile 1 [Mild]
  Interventions: Other: Patient Survey
- Quartile 2 [Moderate]
  Interventions: Other: Patient Survey
- Quartile 3 [Severe]
  Interventions: Other: Patient Survey
- Quartile 4 [Very Severe]
  Interventions: Other: Patient Survey

INTERVENTIONS:
Other: Patient Survey — Participants will answer an online survey and their medical chart information will be gathered to compare responses across disease severity.

SUMMARY:
The purpose of this study is to distribute a questionnaire created for individuals living with chronic obstructive pulmonary disease (COPD) to assess their activities, participation, and healthcare and COPD-related research priorities. The data collected will be compared across diagnosed COPD stages and disease severity to determine the extent to which adults with COPD participate in the listed activities and identify their primary research and healthcare related priorities. The questionnaire was originally developed based on past research then verified by a panel of COPD and participation experts; as well as, individuals living with COPD in the form of focus groups. The questionnaire will now be administered to 200 individuals living COPD (50 in each GOLD stage) at three sites across Montreal where clinical data for each participant will be available. This phase will help establish the reliability of the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD
* English or French speaking
* Patient at one of the three participating sites with medical chart

Exclusion Criteria:

* No diagnosis of COPD by a healthcare professional
* Unable to communicate in English or French
* Unable to provide informed consent
* No medical chart information at one of the three participating sites

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults living with chronic obstructive pulmonary disease (COPD).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-11; Primary Completion 2017-10 (Actual); Study Completion 2018-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Jensen, Ph.D., Principal Investigator — McGill University; Shane N Sweet, Ph.D., Principal Investigator — McGill University
Locations (1):
- Montreal Chest Institute of the McGill University Health Center (MUHC), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Exercise and Respiratory Physiology Laboratory (CERPL) — http://www.mcgill.ca/cerpl/
- See also: Theories and Interventions in Exercise and Health Psychology (TIE) Laboratory — http://exercisepsych.research.mcgill.ca/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 200 participants completed the AHRPQ. Of those, 52 were missing spirometry in medical records, 148 completed with spirometry for Quartile 1-4 analysis [groups], and 130 of the 148 completed spirometry, exacerbation and mMRC for Group A-D analysis.
Groups:
- All Participants: Participants answered an online survey and their medical chart information was gathered to compare responses across disease severity. This was a single arm study.
Period: Overall Study
Arm/Group | All Participants
Started | 200
Completed | 200
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 200
Age, Continuous [Median (Standard Deviation); unit: Years] | 67.5 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants were missing data as data collected was voluntary to provide or the information was not included in their medical charts.
  Participants
    number analyzed (Participants) | 199
    Female | 96
    Male | 103
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Participants were missing data as data collected was voluntary to provide or the information was not included in their medical charts.
  Participants
    Race: number analyzed (Participants) | 193
    Race: Other | 12
    Race: White | 181
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 200
Marital Status [Count of Participants; unit: Participants] — Population: Participants were missing data as data collected was voluntary to provide or the information was not included in their medical charts.
  Participants
    number analyzed (Participants) | 194
    Single/Divorced/Widowed | 86
    Married/Common Law | 108
Education [Count of Participants; unit: Participants] — Population: Participants were missing data as data collected was voluntary to provide or the information was not included in their medical charts.
  Participants
    number analyzed (Participants) | 194
    Full-time/Part-time | 86
    Unemployed/Retired/Disability | 108
Household Income [Count of Participants; unit: Participants] — Population: Participants were missing data as data collected was voluntary to provide or the information was not included in their medical charts.
  Participants
    number analyzed (Participants) | 161
    Under $60,000 | 118
    Above $60,000 | 43
Smoking [Count of Participants; unit: Participants] — Population: Participants were missing data as data collected was voluntary to provide or the information was not included in their medical charts.
  Participants
    number analyzed (Participants) | 193
    Never smoked tobacco | 9
    Ever smoked tobacco | 184
CAT (COPD assessment test) [Count of Participants; unit: Participants] — This questionnaire helps measure the impact COPD is having on well being and daily life. The CAT is an eight-item semantic differential scale from 0 to 5, where 0 is no impact and 5 is extremely impactful. Individuals are asked to rate the impact of 8 items on their COPD disease burden. Their total score is calculated. A score of <10 is representative of lower disease burden; whereas, a score >= 10 is indicative of higher disease burden. Population: Participants were missing data as data collected was voluntary to provide or the information was not included in their medical charts.
  Participants
    score <10 (less than normal burden of disease): number analyzed (Participants) | 197
    score <10 (less than normal burden of disease) | 34
    score ≥10 (higher than normal burden of disease ) | 163
mMRC (Modified-Medical Research Council Questionnaire on breathlessness) [Count of Participants; unit: Participants] — This questionnaire was used to measure participants' breathlessness burden using a single item scale from 0 to 4, where a score of 0-1 indicated mild breathlessness and 2-4 indicated increased breathlessness. Population: Participants were missing data as data collected was voluntary to provide or the information was not included in their medical charts.
  Participants
    number analyzed (Participants) | 196
    0-1 (mild breathlessnes) | 67
    ≥2 (increased breathlessness) | 129
Pulmonary Rehab Attendance [Count of Participants; unit: Participants] — Population: Participants were missing data as data collected was voluntary to provide or the information was not included in their medical charts.
  Participants
    number analyzed (Participants) | 193
    Yes | 81
    No | 112
Myocardial Infarction [Count of Participants; unit: Participants] | 11
Congestive heart failure [Count of Participants; unit: Participants] | 15
Peripheral vascular disease [Count of Participants; unit: Participants] | 7
Cerebrovascular disease [Count of Participants; unit: Participants] | 3
Dementia [Count of Participants; unit: Participants] | 1
Connective tissue disease [Count of Participants; unit: Participants] | 3
Diabetes Mellitus [Count of Participants; unit: Participants] | 18
Chronic kidney disease [Count of Participants; unit: Participants] | 5
Hemiplegia [Count of Participants; unit: Participants] | 0
Cancer [Count of Participants; unit: Participants] | 25
Liver disease [Count of Participants; unit: Participants] | 4
HIV/AIDS [Count of Participants; unit: Participants] | 1
Asthma [Count of Participants; unit: Participants] | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Prioritized Healthcare Topics
Description: Twenty-four healthcare topics were selected once again from a literature and expert panel review, as well as corroborated by individuals living with COPD in five focus groups. Example healthcare topics include: relief of breathlessness; increase maximal amount of exercise individuals living with COPD can do inside and outside their homes; and prevent-lung flare-ups. Participants were asked to indicate their preference of the topics by assigning a percentage of their time, in increments of 10%, to the various healthcare topics, for a total of 100% of their time. For the 24 healthcare topics, individuals could select up to 10 topics (10% times 10 topics, for 100% of their time). The top five topics are presented as the most important topics for the participants and are indicative of areas of focus for future healthcare and research. The top five were presented in accordance to the request from the working group who developed the survey and reviewed the results.
Time Frame: Baseline
Population: Participants answered an online survey and their medical chart information was gathered to compare responses across disease severity. Of the 148 participants, 130 completed the online survey with spirometry & exacerbation and mMRC for Group ABCD analysis.
Measure: Number; unit: participants
Groups:
- Participation Differences by Individuals' Disease Severity: For airflow obstruction, individuals were divided into quartiles based on their FEV1%predicted. (mild, moderate, severe, and very severe)
- Participation Differences by (GOLD) ABCD Classification: Individuals' ABCD classifications were based on the 2017 GOLD guidelines based on modified British Medical Research Council (mMRC) dyspnea scores and 12-month exacerbation history.
- Quartile 1 - Mild Airflow Obstruction: FEV1%predicted range = 65.1-184.8
- Quartile 2 - Moderate Airflow Obstruction: FEV1% predicted range = 48.4-64.3
- Quartile 3 - Severe Airflow Obstruction: FEV1% predicted range = 31.7-46.8
- Quartile 4 - Very Severe Airflow Obstruction: FEV1% predicted range = 14.7-31.5
- Group A - Breathlessness Burden and Exacerbation Risk: FEV1%predicted range = 42.3-69.4
- Group B - Breathlessness Burden and Exacerbation Risk: FEV1% predicted range = 28.0-65.9
- Group C - Breathlessness Burden and Exacerbation Risk: FEV1% predicted range = 27.0-67.0
- Group D - Breathlessness Burden and Exacerbation Risk: FEV1% predicted range = 27.0-67.7
Arm/Group | Participation Differences by Individuals' Disease Severity | Participation Differences by (GOLD) ABCD Classification | Quartile 1 - Mild Airflow Obstruction | Quartile 2 - Moderate Airflow Obstruction | Quartile 3 - Severe Airflow Obstruction | Quartile 4 - Very Severe Airflow Obstruction | Group A - Breathlessness Burden and Exacerbation Risk | Group B - Breathlessness Burden and Exacerbation Risk | Group C - Breathlessness Burden and Exacerbation Risk | Group D - Breathlessness Burden and Exacerbation Risk
Number analyzed (Participants) | 148 | 130 | 37 | 37 | 37 | 37 | 26 | 50 | 14 | 40
participants
  Relief of Breathlessness | 90 | 79 | 23 | 22 | 21 | 24 | 11 | 36 | 5 | 27
  Improve Your Ability to Improve Activities | 79 | 67 | 20 | 22 | 15 | 22 | 12 | 30 | 6 | 19
  Prevent Lung Flare-Ups | 74 | 64 | 18 | 18 | 18 | 20 | 14 | 23 | 7 | 20
  Discuss COPD | 71 | 61 | 18 | 19 | 23 | 11 | 12 | 27 | 6 | 16
  Improve Physical Well-Being | 70 | 62 | 20 | 15 | 17 | 18 | 12 | 26 | 9 | 15
Statistical Analysis 1: Comparison: Participation Differences by Individuals' Disease Severity; Relief of breathlessness; Test type: Other; p = .91, Chi-squared; Chi-squared value= .57
Statistical Analysis 2: Comparison: Participation Differences by Individuals' Disease Severity; Improve your ability to perform activities in and out of your home; Test type: Other; p = .31, Chi-squared; Chi-squared value= 3.56
Statistical Analysis 3: Comparison: Participation Differences by Individuals' Disease Severity; Prevent lung flare-ups; Test type: Other; p = .96, Chi-squared; Chi-squared value=.32
Statistical Analysis 4: Comparison: Participation Differences by Individuals' Disease Severity; Discuss COPD and its progression; Test type: Other; p = .04, Chi-squared; Chi-squared value= 8.09
Statistical Analysis 5: Comparison: Participation Differences by Individuals' Disease Severity; Improve your physical well-being; Test type: Other; p = .70, Chi-squared; Chi-squared value: 1.41
Statistical Analysis 6: Comparison: Participation Differences by (GOLD) ABCD Classification; Relief of breathlessness; Test type: Other; p = .01, Chi-squared; Chi-squared value= 10.81
Statistical Analysis 7: Comparison: Participation Differences by (GOLD) ABCD Classification; Improve your ability to perform activities in and out of your home; Test type: Other; p = .49, Chi-squared; Chi-squared value= 2.41
Statistical Analysis 8: Comparison: Participation Differences by (GOLD) ABCD Classification; Prevent lung flare-ups; Test type: Other; p = .93, Chi-squared; Chi-squared value= .44
Statistical Analysis 9: Comparison: Participation Differences by (GOLD) ABCD Classification; Discuss COPD and its progression; Test type: Other; p = .60, Chi-squared; Chi-squared value= 1.87
Statistical Analysis 10: Comparison: Participation Differences by (GOLD) ABCD Classification; Improve your physical well-being; Test type: Other; p = .31, Chi-squared; Chi-squared value= 3.61

2. Primary Outcome: Number of Participants Who Prioritized Research Topics
Description: Individuals were asked to indicate their research priorities from a list of research topics using a modified willingness-to-pay method (Kawata et al., 2014). The willingness-to-pay method allows individuals to assign preference to various topics by assigning a percentage of funds to the topic. A list of 22 research topics (e.g., to relieve breathlessness in individuals living with COPD, to increase access to lung transplantations) was created for this study through a literature review, expert consultation, and five focus groups with individuals living with COPD (n=23, 27% women). Individuals were asked to assign a percentage of funds, in increments of 10% of funding, to the 22 COPD research topics. Participants could assign anywhere between 10% of funding to 100% of funding to the topics. The top five were presented in accordance to the request from the working group who developed the survey and reviewed the results.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Participation Differences by Individuals' Disease Severity | Participation Differences by (GOLD) ABCD Classification | Quartile 1 - Mild Airflow Obstruction | Quartile 2 - Moderate Airflow Obstruction | Quartile 3 - Severe Airflow Obstruction | Quartile 4 - Very Severe Airflow Obstruction | Group A - Breathlessness Burden and Exacerbation Risk | Group B - Breathlessness Burden and Exacerbation Risk | Group C - Breathlessness Burden and Exacerbation Risk | Group D - Breathlessness Burden and Exacerbation Risk
Number analyzed (Participants) | 148 | 130 | 37 | 37 | 37 | 37 | 26 | 50 | 14 | 40
participants
  To relieve breathlessness in COPD | 113 | 98 | 28 | 29 | 26 | 30 | 20 | 40 | 7 | 31
  To prevent the development of COPD | 85 | 74 | 18 | 26 | 22 | 19 | 15 | 30 | 9 | 20
  To prevent lung flare ups | 74 | 62 | 18 | 18 | 14 | 24 | 14 | 24 | 3 | 21
  To increase the ability to exercise | 70 | 61 | 20 | 14 | 17 | 19 | 11 | 29 | 7 | 14
  To improve maximal amount of exercise | 68 | 57 | 21 | 12 | 15 | 20 | 6 | 29 | 4 | 18
Statistical Analysis 1: Comparison: Participation Differences by Individuals' Disease Severity; To relieve breathlessness in adults living with COPD; Test type: Other; p = .73, Chi-squared; Chi-squared value: 1.31
Statistical Analysis 2: Comparison: Participation Differences by Individuals' Disease Severity; To prevent the development of COPD; Test type: Other; p = .23, Chi-squared; Chi-squared value= 4.28
Statistical Analysis 3: Comparison: Participation Differences by Individuals' Disease Severity; To prevent lung flare-ups in adults living with COPD; Test type: Other; p = .14, Chi-squared; Chi-squared value= 5.51
Statistical Analysis 4: Comparison: Participation Differences by Individuals' Disease Severity; To increase the ability of adults living with COPD to exercise; Test type: Other; p = .52, Chi-squared; Chi-squared value= 2.28
Statistical Analysis 5: Comparison: Participation Differences by Individuals' Disease Severity; To improve the maximal amount of exercise of adults living with COPD in and out of the home; Test type: Other; p = .11, Chi-squared; Chi-squared value= 5.88
Statistical Analysis 6: Comparison: Participation Differences by (GOLD) ABCD Classification; To relieve breathlessness in adults living with COPD; Test type: Other; p = .14, Chi-squared; Chi-squared value= 5.57
Statistical Analysis 7: Comparison: Participation Differences by (GOLD) ABCD Classification; To prevent the development of COPD; Test type: Other; p = .73, Chi-squared; Chi-squared value= 1.29
Statistical Analysis 8: Comparison: Participation Differences by (GOLD) ABCD Classification; To prevent lung flare-ups in adults living with COPD; Test type: Other; p = .20, Chi-squared; Chi-squared value= 4.64
Statistical Analysis 9: Comparison: Participation Differences by (GOLD) ABCD Classification; To increase the ability of adults living with COPD to exercise; Test type: Other; p = .17, Chi-squared; Chi-squared value= 5.02
Statistical Analysis 10: Comparison: Participation Differences by (GOLD) ABCD Classification; To improve the maximal amount of exercise of adults living with COPD in and out of the home; Test type: Other; p = .02, Chi-squared; Chi-square value= 9.97

3. Primary Outcome: Number of Participants Who Were Not Satisfied With Their Participation in Daily and Social Activities
Description: Participants will answer questions about their participation in 26 daily activities, as well as their desire to participate in each of the 26 daily activities. This is a measure of those who indicated they wanted to increase their participation. 10 of the 26 activities and their outcome measures are listed below.
  Activity 1: Walking from one place to another outside of your home on a flat surface.
  Activity 2: Moving from one place to another using motorized transportation.
  Activity 3: Climbing two or more flights of stairs.
  Activity 4: Walking up a hill.
  Activity 5: Participating in regular exercise.
  Activity 6: Walking from one place to another in your home.
  Activity 7: Carrying light objects on a flat surface.
  Activity 8: Carrying heavy objects on a flat surface.
  Activity 9: Carrying-out low intensity physical activities
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Participation Differences by Individuals' Disease Severity | Participation Differences by (GOLD) ABCD Classification | Quartile 1 - Mild Airflow Obstruction | Quartile 2 - Moderate Airflow Obstruction | Quartile 3 - Severe Airflow Obstruction | Quartile 4 - Very Severe Airflow Obstruction | Group A - Breathlessness Burden and Exacerbation Risk | Group B - Breathlessness Burden and Exacerbation Risk | Group C - Breathlessness Burden and Exacerbation Risk | Group D - Breathlessness Burden and Exacerbation Risk
Number analyzed (Participants) | 148 | 130 | 37 | 37 | 37 | 37 | 26 | 50 | 14 | 40
participants
  Activity 1 | 108 | 83 | 8 | 27 | 30 | 43 | 8 | 38 | 7 | 30
  Activity 2 | 17 | 25 | 5 | 3 | 3 | 6 | 15 | 2 | 0 | 8
  Activity 3 | 114 | 101 | 24 | 27 | 22 | 41 | 12 | 30 | 21 | 38
  Activity 4 | 142 | 107 | 24 | 41 | 39 | 38 | 19 | 44 | 0 | 44
  Activity 5 | 117 | 87 | 22 | 22 | 32 | 41 | 8 | 44 | 7 | 28
  Activity 6 | 3 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
  Activity 7 | 19 | 15 | 5 | 3 | 3 | 8 | 4 | 6 | 0 | 5
  Activity 8 | 99 | 86 | 11 | 22 | 28 | 38 | 7 | 27 | 14 | 38
  Activity 9 | 30 | 28 | 5 | 3 | 3 | 19 | 8 | 8 | 7 | 5
  Activity 10 | 90 | 71 | 5 | 17 | 30 | 38 | 0 | 24 | 14 | 33
Statistical Analysis 1: Comparison: Participation Differences by Individuals' Disease Severity; Activity 1: Walking from one place to another outside of your home on a flat surface; Test type: Other; p = .05, Chi-squared; Chi squared value= 17.20
Statistical Analysis 2: Comparison: Participation Differences by Individuals' Disease Severity; Activity 2: Moving from one place to another using motorized transportation; Test type: Other; p = .87, Chi-squared; Chi-squared value= 4.56
Statistical Analysis 3: Comparison: Participation Differences by Individuals' Disease Severity; Activity 3: Climbing two or more flights of stairs; Test type: Other; p = .65, Chi-squared; Chi-squared value= 6.85
Statistical Analysis 4: Comparison: Participation Differences by Individuals' Disease Severity; Activity 4: Walking up a hill; Test type: Other; p = .35, Chi-squared; Chi-squared value= 10.00
Statistical Analysis 5: Comparison: Participation Differences by Individuals' Disease Severity; Activity 5: Participating in regular exercise requiring physical effort, to maintain or improve health or fitness; Test type: Other; p = .03, Chi-squared; Chi-squared value= 18.75
Statistical Analysis 6: Comparison: Participation Differences by (GOLD) ABCD Classification; Activity 1: Walking from one place to another outside of your home on a flat surface; Test type: Other; p = .00, Chi-squared; Chi-squared value= 35.52
Statistical Analysis 7: Comparison: Participation Differences by (GOLD) ABCD Classification; Activity 2: Moving from one place to another using motorized transportation; Test type: Other; p = .33, Chi-squared; Chi-squared value= 10.23
Statistical Analysis 8: Comparison: Participation Differences by (GOLD) ABCD Classification; Activity 3: Climbing two or more flights of stairs; Test type: Other; p = .00, Chi-squared; Chi-squared value= 23.94
Statistical Analysis 9: Comparison: Participation Differences by (GOLD) ABCD Classification; Activity 4: Walking up a hill; Test type: Other; p = .01, Chi-squared; Chi-squared value= 22.80
Statistical Analysis 10: Comparison: Participation Differences by (GOLD) ABCD Classification; Activity 5: Participating in regular exercise requiring physical effort, to maintain or improve health or fitness; Test type: Other; p = .02, Chi-squared; Chi-squared value= 20.43

4. Secondary Outcome: Forced Expiratory Volume in 1-sec (FEV1)
Description: Individuals forced expiratory volume in 1-sec (FEV1) as assessed by spirometry
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percent predicted
Groups:
- Participation Differences by (GOLD) ABCD: Individuals' ABCD classifications were based on the 2017 GOLD guidelines based on modified British Medical Research Council (mMRC) dyspnea scores and 12-month exacerbation history.
Arm/Group | Participation Differences by Individuals' Disease Severity | Participation Differences by (GOLD) ABCD | Quartile 1 - Mild Airflow Obstruction | Quartile 2 - Moderate Airflow Obstruction | Quartile 3 - Severe Airflow Obstruction | Quartile 4 - Very Severe Airflow Obstruction | Group A - Breathlessness Burden and Exacerbation Risk | Group B - Breathlessness Burden and Exacerbation Risk | Group C - Breathlessness Burden and Exacerbation Risk | Group D - Breathlessness Burden and Exacerbation Risk
Number analyzed (Participants) | 148 | 130 | 37 | 37 | 37 | 37 | 26 | 50 | 14 | 40
percent predicted | 49.6 (23.2) | 48.5 (20.7) | 79.0 (21.5) | 55.6 (5.5) | 38.5 (4.8) | 25.2 (4.5) | 66.0 (20.2) | 47.1 (17.9) | 50.8 (20.3) | 37.8 (17.0)
Statistical Analysis 1: Comparison: Participation Differences by Individuals' Disease Severity; Test type: Other; p = .00, Kruskal-Wallis; Non-parametric led to equal variance (levene's test) which couldn't be assumed, independent samples were taken (Kruskal-Wallis); F(3,144)=137.82

5. Secondary Outcome: FEV1/FVC
Description: Individuals FEV1-to-forced vital capacity (FVC) ratio
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Measured ratio
Arm/Group | Participation Differences by Individuals' Disease Severity | Participation Differences by (GOLD) ABCD | Quartile 1 - Mild Airflow Obstruction | Quartile 2 - Moderate Airflow Obstruction | Quartile 3 - Severe Airflow Obstruction | Quartile 4 - Very Severe Airflow Obstruction | Group A - Breathlessness Burden and Exacerbation Risk | Group B - Breathlessness Burden and Exacerbation Risk | Group C - Breathlessness Burden and Exacerbation Risk | Group D - Breathlessness Burden and Exacerbation Risk
Number analyzed (Participants) | 148 | 130 | 37 | 37 | 37 | 37 | 26 | 50 | 14 | 40
Measured ratio | 49.1 (11.8) | 49.0 (11.9) | 60.5 (8.5) | 53.8 (8.5) | 44.1 (8.9) | 38.1 (7.9) | 58.1 (7.3) | 47.9 (11.2) | 49.1 (12.8) | 44.5 (12.0)
Statistical Analysis 1: Comparison: Participation Differences by Individuals' Disease Severity; Test type: Other; p = .000, ANOVA; Factorial ANOVA used because variance could be assumed; F(3,144)=55.89 Partial ETA squared (effect size)=0.54

6. Secondary Outcome: Modified Medical Research Council Questionnaire on Breathlessness
Description: Self-reported intensity of activity related breathlessness as assessed by the modified Medical Research Council (mMRC) dyspnea scale (0-4). This questionnaire was used to measure participants' breathlessness burden using a single item scale from 0 to 4, where a score of 0-1 indicated mild breathlessness and 2-4 indicated increased breathlessness.
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Participation Differences by Individuals' Disease Severity | Participation Differences by (GOLD) ABCD | Quartile 1 - Mild Airflow Obstruction | Quartile 2 - Moderate Airflow Obstruction | Quartile 3 - Severe Airflow Obstruction | Quartile 4 - Very Severe Airflow Obstruction | Group A - Breathlessness Burden and Exacerbation Risk | Group B - Breathlessness Burden and Exacerbation Risk | Group C - Breathlessness Burden and Exacerbation Risk | Group D - Breathlessness Burden and Exacerbation Risk
Number analyzed (Participants) | 148 | 130 | 37 | 37 | 37 | 37 | 26 | 50 | 14 | 40
participants
  mMRC 0-1 | 45 | 40 | 20 | 15 | 7 | 3 | 26 | 0 | 14 | 0
  mMRC ≥2 | 101 | 90 | 15 | 22 | 30 | 34 | 0 | 50 | 0 | 40
  Data missing | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Participation Differences by Individuals' Disease Severity; Test type: Other; p = .00, ANOVA; One-way ANOVA; F(3,142)=7.61

7. Secondary Outcome: COPD Assessment Test
Description: This questionnaire measure the impact COPD is having on well being and daily life. The CAT is an eight-item semantic differential scale from 0 to 5, where 0 is no impact and 5 is extremely impactful. Items include: I never cough| I cough all the time, I have no phlegm (mucus) in my chest at all | My chest is completely full of phlegm (mucus), My chest does not feel tight at all | My chest feels very tight, When I walk up a hill or one flight of stairs, I am not breathless | When I walk up a hill or one flight of stairs, I am very breathless, I am not limited doing any activities at home| I am very limited doing activities at home, I am confident leaving my home despite my lung condition| I am not at all confident leaving my home because of my lung condition, I sleep soundly | I don't sleep soundly because of my lung condition, I have lots of energy I have no energy at all. Participants' scores were totaled and a score of ≥ 10 indicated higher than normal burden of disease.
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Participation Differences by Individuals' Disease Severity | Participation Differences by (GOLD) ABCD | Quartile 1 - Mild Airflow Obstruction | Quartile 2 - Moderate Airflow Obstruction | Quartile 3 - Severe Airflow Obstruction | Quartile 4 - Very Severe Airflow Obstruction | Group A - Breathlessness Burden and Exacerbation Risk | Group B - Breathlessness Burden and Exacerbation Risk | Group C - Breathlessness Burden and Exacerbation Risk | Group D - Breathlessness Burden and Exacerbation Risk
Number analyzed (Participants) | 148 | 130 | 37 | 37 | 37 | 37 | 26 | 50 | 14 | 40
participants
  CAT <10 | 24 | 22 | 10 | 5 | 6 | 3 | 8 | 6 | 5 | 3
  CAT ≥10 | 122 | 107 | 26 | 32 | 30 | 34 | 18 | 44 | 9 | 36
  Data missing | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Participation Differences by Individuals' Disease Severity; Test type: Other; p = .31, ANOVA; One-way ANOVA; F(3,142)=1.21

8. Secondary Outcome: Godin Leisure Time Physical Activity Questionnaire
Description: Self-reported physical activity levels measured in length of bouts over the previous 7 days to determine physical activity frequency.
Time Frame: Baseline
Population: Missing data n=8 for differences by individuals' disease severity and n=4 for differences by (GOLD) ABCD
Measure: Mean (Standard Deviation); unit: Total minutes of Moderate to Vigorous PA
Groups:
- Quartile 1- Mild Airflow Obstruction: FEV1% predicted range: 65.1-184.8
- Quartile 2 - Moderate Airflow Obstruction: FEV1% predicted range: 48.4-64.3
- Quartile 3 - Severe Airflow Obstruction: FEV1% predicted range: 31.7-46.8
- Quartile 4 - Very Severe Airflow Obstruction: FEV1% predicted range: 14.7-31.5
- Group A - Breathlessness Burden and Exacerbation Risk: FEV1% predicted range: 42.3-69.4
- Group B - Breathlessness Burden and Exacerbation Risk: FEV1% predicted range:28.0-65.9
- Group C - Breathlessness Burden and Exacerbation Risk; Group D - Breathlessness Burden and Exacerbation Risk: FEV1% predicted range:27.0-67.0
Arm/Group | Participation Differences by Individuals' Disease Severity | Participation Differences by (GOLD) ABCD | Quartile 1- Mild Airflow Obstruction | Quartile 2 - Moderate Airflow Obstruction | Quartile 3 - Severe Airflow Obstruction | Quartile 4 - Very Severe Airflow Obstruction | Group A - Breathlessness Burden and Exacerbation Risk | Group B - Breathlessness Burden and Exacerbation Risk | Group C - Breathlessness Burden and Exacerbation Risk | Group D - Breathlessness Burden and Exacerbation Risk
Number analyzed (Participants) | 140 | 126 | 34 | 35 | 36 | 35 | 23 | 50 | 14 | 39
Total minutes of Moderate to Vigorous PA | 74.64 (138.59) | 101.86 (194.49) | 100.29 (170.08) | 117.06 (175.61) | 42.78 (90.57) | 40.06 (79.70) | 166.52 (204.52) | 33.38 (76.05) | 138.57 (149.35) | 39.10 (73.21)
Statistical Analysis 1: Comparison: Participation Differences by Individuals' Disease Severity; Test type: Other; p = .04, Kruskal-Wallis; Non-parametric independent sample Kruskal-Wallis test (failed variance assumed; F(3,139)=8.09

9. Secondary Outcome: Satisfaction of Life Questionnaire
Description: This 5 item questionnaire was used to measure participants' level of life satisfaction. The higher the score, the higher the sense of life satisfaction. A score from 5-9 indicated extremely dissatisfied, 10-14 is dissatisfied, 15-19 indicated slightly below average life satisfaction. 20-24 is the average score, 25-29 is a high score indicative of higher life satisfaction and a score between 30-35 is a very high score and represent very high life satisfaction.
Time Frame: Baseline
Population: Missing data n=6 for differences by individuals' disease severity and n=6 for differences by (GOLD) ABCD
Measure: Mean (Standard Deviation); unit: total score on a scale
Groups:
- Quartile 4 - Very Severe Airflow Obstruction: Quartile 4 - Very Severe Airflow Obstruction
Arm/Group | Participation Differences by Individuals' Disease Severity | Participation Differences by (GOLD) ABCD | Quartile 1- Mild Airflow Obstruction | Quartile 2 - Moderate Airflow Obstruction | Quartile 3 - Severe Airflow Obstruction | Quartile 4 - Very Severe Airflow Obstruction | Group A - Breathlessness Burden and Exacerbation Risk | Group B - Breathlessness Burden and Exacerbation Risk | Group C - Breathlessness Burden and Exacerbation Risk | Group D - Breathlessness Burden and Exacerbation Risk
Number analyzed (Participants) | 142 | 124 | 35 | 33 | 37 | 37 | 26 | 46 | 12 | 40
total score on a scale | 18.62 (8.16) | 18.38 (8.14) | 22.51 (7.78) | 20.94 (7.68) | 16.35 (7.23) | 15.1 (7.87) | 22.50 (6.83) | 17.33 (8.10) | 21.67 (6.73) | 15.95 (8.26)
Statistical Analysis 1: Comparison: Participation Differences by Individuals' Disease Severity; Test type: Other; p = .00, ANOVA; One-way ANOVA; F(3,143)=8.01

10. Secondary Outcome: Number of Participants With Exacerbations Due to COPD in the Preceding 12 Months
Description: An exacerbation was defined as a change in medication due to a COPD exacerbation (i.e., the prescription of prednisone or a medical action plan) as indicated in the medical chart or hospital admission due to a COPD exacerbation.
Time Frame: baseline
Measure: Number; unit: participants
Arm/Group | Participation Differences by Individuals' Disease Severity | Participation Differences by (GOLD) ABCD | Quartile 1- Mild Airflow Obstruction | Quartile 2 - Moderate Airflow Obstruction | Quartile 3 - Severe Airflow Obstruction | Quartile 4 - Very Severe Airflow Obstruction | Group A - Breathlessness Burden and Exacerbation Risk | Group B - Breathlessness Burden and Exacerbation Risk | Group C - Breathlessness Burden and Exacerbation Risk | Group D - Breathlessness Burden and Exacerbation Risk
Number analyzed (Participants) | 148 | 130 | 37 | 37 | 37 | 37 | 26 | 50 | 14 | 40
participants
  Number of participants with 0-1 exacerbations | 92 | 76 | 30 | 27 | 19 | 16 | 26 | 50 | 0 | 0
  Number of participants with 2+ or 1 exacerbations leading to hospital admission | 56 | 54 | 7 | 10 | 18 | 21 | 0 | 0 | 14 | 40

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not assessed.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/22/NCT02970422/ICF_000.pdf
  • Study Protocol (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/22/NCT02970422/Prot_001.pdf
  • Statistical Analysis Plan (2019-09-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT02970422/SAP_002.pdf